CLINICAL TRIAL: NCT02481037
Title: Primary Care Pathway for Childhood Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Alberta Health Services, Calgary (Other); Health Quality Council of Alberta (HQCA) (Unknown); University of Calgary (Other); Ottawa Hospital Research Institute (Other); TELUS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201400389
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Embedding a primary care clinical pathway for managing childhood asthma into clinicians' electronic medical record (EMR) to facilitate practitioners utilizing best-evidence; training these practices' chronic disease management (CDM) professionals to provide asthma education to children with asthma and their parents; and clinicians receiving an EMR embedded dashboard.
  Interventions: Other: Primary care clinical pathway; Other: Asthma education; Other: EMR embedded dashboard
- Control group (No Intervention): Practice will continue with routine care. Control group will be offered the intervention at study completion, if successful.

INTERVENTIONS:
Other: Primary care clinical pathway — Installing a primary care clinical pathway for managing childhood asthma into clinicians' electronic medical record (EMR) to facilitate the use of best-evidence by practitioners.
  Arms: Intervention group
Other: Asthma education — Physicians will receive web-based education through an interactive learning module regarding best management for childhood asthma and use of the primary care clinical pathway. Chronic disease management (CDM) health professionals in practices will attend asthma education sessions delivered by an asthma educator. This training will be then used by the CDM professional to provide targeted and timely asthma education to parents and children with asthma.
  Arms: Intervention group
Other: EMR embedded dashboard — An EMR embedded dashboard will deliver real-time feedback to clinicians.
  Arms: Intervention group

SUMMARY:
At least half of children with asthma have poor disease control, which can result in complications requiring emergency treatment and hospitalization. As asthma is one of the most common reasons for children to visit emergency departments (ED) and be hospitalized, this disease places a heavy burden on the health care system and families. While there is strong evidence that timely treatment with preventative therapies can substantially improve asthma control, reduce sudden worsening of symptoms, and lower rates of ED visits and hospitalizations, a significant proportion of children do not receive these therapies.

The purpose of this study is to improve the prescription and use of evidenced-based preventative therapies for children with asthma with the goal to significantly improve their disease control and quality of life, while reducing unnecessary ED visits and hospitalizations. The investigators will achieve this by: i) installing a primary care clinical pathway for managing childhood asthma into clinicians' electronic medical record (EMR) to facilitate the use of best-evidence by practitioners, and ii) training chronic disease management (CDM) health professionals to provide targeted and timely asthma education to parents and children with asthma. The investigators will test this pathway and education project in a representative sample of 22 Alberta primary care practices, using a pragmatic cluster controlled trial methodology.

ELIGIBILITY:
Inclusion Criteria:

* Validated diagnosis of asthma according to CPCSSN validated definition

Exclusion Criteria:

* Children under 1 and over 17 years of age
* Children of parents who have opted out of CPCSSN data collection
* Children with validated asthma who have not attended practices in the last 2 years, or have not received bronchodilator therapy in the last 12 months

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Prescription of evidenced-based preventative therapies | 12 months after receiving intervention
  The proportion of symptomatic children with asthma in the baseline and follow-up periods (separate calculations) who are appropriately treated with a preventer will be the primary outcome. The denominator will be the number of children who meet the case definition of asthma and receive at least one prescription for an inhaled short-acting beta-agonist (e.g. salbutamol) during the applicable time period. The numerator will be, of these children, the number who receive a prescription for inhaled corticosteroid, montelukast, a combined inhaled long-acting beta agonist and corticosteroid, or some combination of these three drugs in the same time period.

SECONDARY OUTCOMES:
Dispensed preventative therapies | 12 months after receiving intervention
  The proportion of applicable children in baseline and follow-up periods who are appropriately dispensed a preventer by a pharmacy will highlight if there is a significant gap between prescriptions given and filled. The denominator will be the same as for the primary outcome but the numerator will be the number of these children who are dispensed one or more preventer medications from newly available Pharmaceutical Information Network (PIN) data.
Emergency department visits and hospitalizations for asthma | 12 months after receiving intervention
  The number of asthma emergency department visits or hospitalizations (ICD10 J45 or J46) per child who meets the case definition of asthma during each time period, a measure of health care use.
Electronic Medical Record (EMR) data | 12 months after receiving intervention
  The research team has worked with TELUS to develop and validate a case definition and case finding algorithm for identifying children with asthma in practices. The TELUS EMR data will provide, for all eligible children, individual categorical and continuous patient level data such as patient demographics, ICD9 codes and medication prescriptions, and for children evaluated in practices randomized to the pathway group, asthma phenotype and provision of asthma action plans.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cave, FCFP, FRCGP, Principal Investigator — Department of Family Medicine, University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potestio ML, Sharpe H, Johnson DW, Grimshaw JM, Faris P, Duan QM, Pow J, Cave A. A cluster randomized controlled trial of an electronic medical record-based pathway for pediatric asthma in primary care in Alberta. CMAJ. 2025 Nov 23;197(40):E1330-E1336. doi: 10.1503/cmaj.241694. PMID 41285460
- [Derived] Sharpe H, Potestio M, Cave A, Johnson DW, Scott SD. Facilitators and barriers to the implementation of the Primary Care Asthma Paediatric Pathway: a qualitative analysis. BMJ Open. 2022 May 12;12(5):e058950. doi: 10.1136/bmjopen-2021-058950. PMID 35551084
- [Derived] Cave AJ, Sharpe H, Anselmo M, Befus AD, Currie G, Davey C, Drummond N, Graham J, Green LA, Grimshaw J, Kam K, Manca DP, Nettel-Aguirre A, Potestio ML, Rowe BH, Scott SD, Williamson T, Johnson DW. Primary Care Pathway for Childhood Asthma: Protocol for a Randomized Cluster-Controlled Trial. JMIR Res Protoc. 2016 Mar 8;5(1):e37. doi: 10.2196/resprot.5261. PMID 26955763